CLINICAL TRIAL: NCT00001296
Title: A Randomized Phase III Trial of Hyperthermic Isolated Limb Perfusion With Melphalan, Tumor Necrosis Factor, and Interferon-Gamma in Patients With Locally Advanced Extremity Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920105; 92-C-0105
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Melanoma
Keywords: Interferon-Gamma; Isolated Limb Perfusion; Melanoma; Melphalan; TNF
MeSH Terms: conditions — Melanoma | interventions — Melphalan; Tumor Necrosis Factor-alpha; Interferon-gamma

INTERVENTIONS:
Drug: melphalan
Drug: tumor necrosis factor
Drug: interferon-gamma
Procedure: hyperthermic isolated limb perfusion

SUMMARY:
Randomized study. Initially, 3 patients will be entered on Arm I as a pilot feasibility study and to standardize the technical aspects of the study. Subsequently, all patients are randomized to Arms I and II.

Arm I: Regional Hyperthermia plus Regional Single-Agent Chemotherapy. Hyperthermic intravenous limb perfusion, HILP; plus Melphalan, L-PAM, NSC-8806.

Arm II: Regional Hyperthermia plus Regional Single-Agent Chemotherapy and Biological Response Modifier Therapy. HILP as in Arm I; plus L-PAM; and Tumor Necrosis Factor (Knoll), TNF, NSC-635257; Interferon gamma (Genentech), IFN-G, NSC-600662.

DETAILED DESCRIPTION:
Patients with locally advanced melanoma confined to an extremity (Stage IIIA or Stage IIIAB) will be treated in a randomized Phase III study with hyperthermic isolated limb perfusion. One arm of the study will be a standard 60 minute perfusion with melphalan as a single agent. The second arm of the study will combine melphalan, tumor necrosis factor, and interferon-gamma in the isolated limb perfusion reproducing a regimen shown to have 100% response rates in a Phase II European trial. Patients will be followed for local response rates, duration of response, treatment toxicity, and disease-free survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Biopsy-proven Stage IIIA or IIIAB melanoma (M.D. Anderson staging system) of an extremity, as follows:

Advanced local disease indicated by 2 or more satellite or in-transit metastases.

Lower limb regional metastases must be distal to the apex of the femoral triangle except inguinal lymph node metastases.

Upper limb regional metastases must be distal to the deltoid insertion except axillary lymph node metastases.

No evidence of systemic disease outside the involved extremity.

Recurrent disease subsequent to prior successful limb perfusion allowed.

Bidimensional directly measurable dermal or subcutaneous lesion required.

PRIOR/CONCURRENT THERAPY:

No prior isolated limb perfusion.

Biologic Therapy: At least 1 month since Biologic Therapy.

At least 3 months since regional therapy of the extremity.

Chemotherapy: At least 1 month since chemotherap.y

At least 3 months since regional therapy of the extremity.

Endocrine Therapy: Not specified.

Radiotherapy: At least 1 month since radiotherapy.

Surgery: Not specified.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0 or 1.

Hematopoietic: Platelets greater than 150,000.

Hepatic: Bilirubin less than 1.5 mg/dl; Coagulation profile normal.

Renal: Creatinine less than 2.0 mg/dl.

Cardiovascular: No evidence of peripheral vascular disease, e.g.:

No history of claudication.

OTHER:

HIV negative.

No pregnant or nursing women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122
Dates: Start 1992-02; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Karakousis CP, Choe KJ, Holyoke ED. Biologic behavior and treatment of intransit metastasis of melanoma. Surg Gynecol Obstet. 1980 Jan;150(1):29-32. PMID 7350699